CLINICAL TRIAL: NCT04340934
Title: The Use of REZUM System in Chinese Male Patients With Lower Urinary Tract Symptom Secondary to Benign Prostate Enlargement
Brief Title: The Use of REZUM System in Chinese Male Patients With LUTS Secondary to Benign Prostate Enlargement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2019.662
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of REZUM system (Experimental): Surgery of benign prostatic hyperplasia by REZUM system
  Interventions: Device: REZUM system

INTERVENTIONS:
Device: REZUM system — Rezūm is a system uses water steam energy to remove the particular part of the prostate that enlarges and causes symptoms due to BPH. Rezum involves a radiofrequency (RF) generator system and an endoscopic device that is introduced into the body via the urethra.

SUMMARY:
Men with enlarged prostates commonly experience lower urinary tract symptoms and may go on to develop complications such as acute urinary retention (AUR). Surgery is the standard treatment option required to remove the enlarged prostates and to rectify such complications. Transurethral resection of prostate (TURP) was first performed over 80 years ago and is still regarded as the "gold standard" for the treatment of benign prostatic enlargement (BPE) in prostates between 30 and 80ml. While TURP results in an improvement in symptoms, perioperative morbidity and long-term complications can include postoperative bleeding, urinary retention, incontinence, urethral strictures, erectile dysfunction, and ejaculatory dysfunction. Rezūm is a system uses water steam energy to remove the particular part of the prostate that enlarges and causes symptoms due to BPH. Rezum involves a radiofrequency (RF) generator system and an endoscopic device that is introduced into the body via the urethra. Radiofrequency energy from the generator will heat up a controlled amount of water inside the system and converting the water into vapour or steam. The thermal energy created outside the body is delivered into the prostate tissue through the tiny needle at the tip of the endoscopic device. Small amount of steam will then be injected into the tissue and energy will be released during the conversion of steam to water. The energy will heat up the prostate tissue and result in gradually removal of the targeted obstructive prostate tissue. The treatment procedure takes approximately 3-7 minutes and can be performed as day surgery. No radiofrequency energy is delivered into the body, other than the prostate. Throughout the procedure normal saline (salty water) is running into the urethra through the scope to help ensure better views and to prevent the urethra from overheating. Voiding symptom will gradually improve after the procedure. From clinical study based in Caucasian population, patients had improved urinary flow rate by on average 50% and also improvement in quality of life scores. The treatment results could last for at least 4 years. However, information regarding the use of Rezum in Chinese and Asian is lacking. This study is proposed to evaluate the efficacy and safety of Rezum in our population.

DETAILED DESCRIPTION:
Benign prostatic enlargement (BPE) is a non-malignant growth of the prostate gland that can lead to a range of lower urinary tract symptoms (LUTS), and in some cases eventually leading to retention of urine. In patients failing to wean off catheter after retention of urine due to BPE, surgical intervention is the standard treatment.

Surgical intervention options have evolved from electrosurgical resection to the use of lasers for enucleation and ablation [1]. Transurethral resection of prostate (TURP) was first performed over 80 years ago and is still regarded as the "gold standard" for the treatment of BPE in prostates between 30 and 80ml [2]. While TURP results in a statistically significant improvement in symptoms score and and maximum urinary flow rate (Qmax), perioperative morbidity and long-term complications can include postoperative bleeding, urinary retention, incontinence, urethral strictures, erectile dysfunction, and ejaculatory dysfunction [3].

Rezum system use the principle of thermodynamic principle of convective energy transfer, which is different to other conductive heat transfer techniques like transurethral microwave therapy or transurethral needle ablation. [4] In the Rezum system, radiofrequency power is used to create thermal energy in the form of water vapor, which in turn deposits the stored thermal energy during the change from steam phase to liquid after injected into the prostatic tissue. The Rezum system contained a generator with a radiofrequency power supply to create water vapor from sterile water and a single-use transurethral delivery device. The tip of the delivery device contains an 18-gauge needle where 12 small emitter holes spaced circumferentially for dispersion of water vapor into the targeted prostatic tissue. The injection is at a pressure slightly higher than interstitial pressure. Due to the convective properties of water vapor, the injected steam will disperse rapidly and homogenously through the tissue and releases stored thermal energy into prostatic tissue. The released thermal energy will cause tissue necrosis. The most important character of the treatment is when the transition zone is treated, its energy will only deposit within the zonal anatomy of the prostate. Studies by histologic and MRI imaging had shown that after treatment, the thermal lesions were only limited to the transition zone without extension to the peripheral zone, bladder, rectum or striated urinary sphincter [5,6]. It was shown that 6 mo after treatment the total prostate volume was reduced by 28.9% and the resolution of thermal lesions as determined with Gadolini- um-enhanced magnetic resonance imaging was almost complete. [6] A small pilot study had shown that Rezum could provide safe and effective treatment upto one year for men with LUTS due to BPE. [7] In the first multicentre, randomised, controlled study 197 men were enrolled and randomised in a 2:1 ratio to treatment with the Rezum system or control. [8] The sham procedure (control) was rigid cystoscopy with imitated treatment sounds. The primary efficacy end point was met at 3 months with relief of symptoms measured by a change in International prostate symptom score (IPSS) of 50% for the treatment arm compared to 20% for the control group (p < 0.0001). In the thermal treatment arm, the maximal uroflow rate increased significantly by 67% from 9.9 ml/s to 16.1 ml/s (p < 0.0001) after 3 months. The clinical beneficial outcome was sustained throughout the study period with an improvement of 54% at the 12-mo follow up. In the latest updated report on the 4-year outcome, the improvement in voiding (as measured by IPSS and uroflowmetry) was sustained to 4 years with surgical retreatment rate of only 4.4%. [9] Therefore, Rezum was proven to be an effective treatment for BPH.

However, all studies focused on the application of Rezum in patients with LUTS are from Caucasian population. Therefore, in this study, investigator plan to evaluate the feasibility and safety of Rezum in the management of Chinese male patients with LUTS secondary to BPE. This could provide information on the tolerability and effectiveness of the treatment in local population.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 50 - 80 years
* clinically indicated for surgical treatment

Exclusion Criteria:

* Patients with active urinary tract infection or in retention of urine
* Patients with bleeding disorder or on anti-coagulation
* Patients with bladder pathology including bladder stone and bladder cancer
* Patients with urethral stricture
* Patients with neurogenic bladder and/or sphincter abnormalities
* Patients with previous nonpharmacological prostate treatment, Prostate cancer
* Fail to give informed consent

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 3 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Changes in International Prostate Symptom Score (IPSS) at 6 months after treatment | at baseline, 6 months after study intervention
  IPSS score ranging from 0-35 (the higher the worse)

SECONDARY OUTCOMES:
Complications rate | 30 days after study intervention
  Complications rate after study intervention
Post-op total score in International Prostate Symptom Score (IPSS) | At 3 months, 6 months and 12 months after study intervention
  Change in total score of IPSS, score ranging from 0-35 (the higher the worse)
Post-op quality of life score | At 3 months, 6 months and 12 months after study intervention
  Change in quality of life assessed by change in International Prostate QOL score (ranges from 0 to 6, the higher the worse)
Post-op International Index of Erectile Function 5 (IIEF-5) score | At 3 months, 6 months and 12 months after study intervention
  Change in total score of International Index of Erectile Function 5 score (ranges from 0 to 25)
Post-op Overactive bladder symptom score (OABSS) score | At 3 months, 6 months and 12 months after study intervention
  Change in total score of Overactive Bladder Symptom Score (ranges from 0 - 15, the higher the worse)
Post-op pain score | Day 0, on the day of study intervention
  Post-treatment pain score ranges from 0 to 10
Change in voiding function in uroflowmetry | At baseline, 3 months, 6 months and 12 months after study intervention
  It is assessed by maximum flow rate in uroflowmetry
Change in urodynamic | At baseline, 3 months, 6 months and 12 months after study intervention
  Change in urodynamic function assessed by flowrate
Change in prostate size | At baseline, 3 months, 6 months and 12 months after study intervention
  Prostate size is assessed by transrectal ultrasound of prostate

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stepanova LA. Comparative evaluation of two methods of calculating zooplankton production exemplified on the Lake Il'men population. Sov J Ecol. 1974 Sep;4(6):476-82. No abstract available. PMID 4445912
- [Background] Gratzke C, Bachmann A, Descazeaud A, Drake MJ, Madersbacher S, Mamoulakis C, Oelke M, Tikkinen KAO, Gravas S. EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. Eur Urol. 2015 Jun;67(6):1099-1109. doi: 10.1016/j.eururo.2014.12.038. Epub 2015 Jan 19. PMID 25613154
- [Background] Rassweiler J, Teber D, Kuntz R, Hofmann R. Complications of transurethral resection of the prostate (TURP)--incidence, management, and prevention. Eur Urol. 2006 Nov;50(5):969-79; discussion 980. doi: 10.1016/j.eururo.2005.12.042. Epub 2006 Jan 30. PMID 16469429
- [Background] Magistro G, Chapple CR, Elhilali M, Gilling P, McVary KT, Roehrborn CG, Stief CG, Woo HH, Gratzke C. Emerging Minimally Invasive Treatment Options for Male Lower Urinary Tract Symptoms. Eur Urol. 2017 Dec;72(6):986-997. doi: 10.1016/j.eururo.2017.07.005. Epub 2017 Jul 19. PMID 28734706
- [Background] Dixon CM, Rijo Cedano E, Mynderse LA, Larson TR. Transurethral convective water vapor as a treatment for lower urinary tract symptomatology due to benign prostatic hyperplasia using the Rezum((R)) system: evaluation of acute ablative capabilities in the human prostate. Res Rep Urol. 2015 Jan 30;7:13-8. doi: 10.2147/RRU.S74040. eCollection 2015. PMID 25674555
- [Background] Mynderse LA, Hanson D, Robb RA, Pacik D, Vit V, Varga G, Wagrell L, Tornblom M, Cedano ER, Woodrum DA, Dixon CM, Larson TR. Rezum System Water Vapor Treatment for Lower Urinary Tract Symptoms/Benign Prostatic Hyperplasia: Validation of Convective Thermal Energy Transfer and Characterization With Magnetic Resonance Imaging and 3-Dimensional Renderings. Urology. 2015 Jul;86(1):122-7. doi: 10.1016/j.urology.2015.03.021. Epub 2015 May 16. PMID 25987496
- [Background] Dixon C, Cedano ER, Pacik D, Vit V, Varga G, Wagrell L, Tornblom M, Mynderse L, Larson T. Efficacy and Safety of Rezum System Water Vapor Treatment for Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. Urology. 2015 Nov;86(5):1042-7. doi: 10.1016/j.urology.2015.05.046. Epub 2015 Jul 26. PMID 26216644
- [Background] McVary KT, Gange SN, Gittelman MC, Goldberg KA, Patel K, Shore ND, Levin RM, Rousseau M, Beahrs JR, Kaminetsky J, Cowan BE, Cantrill CH, Mynderse LA, Ulchaker JC, Larson TR, Dixon CM, Roehrborn CG. Minimally Invasive Prostate Convective Water Vapor Energy Ablation: A Multicenter, Randomized, Controlled Study for the Treatment of Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2016 May;195(5):1529-1538. doi: 10.1016/j.juro.2015.10.181. Epub 2015 Nov 22. PMID 26614889
- [Background] McVary KT, Rogers T, Roehrborn CG. Rezum Water Vapor Thermal Therapy for Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia: 4-Year Results From Randomized Controlled Study. Urology. 2019 Apr;126:171-179. doi: 10.1016/j.urology.2018.12.041. Epub 2019 Jan 21. PMID 30677455
- [Background] Cantrill CH, Zorn KC, Elterman DS, Gonzalez RR. The Rezum system - a minimally invasive water vapor thermal therapy for obstructive benign prostatic hyperplasia. Can J Urol. 2019 Jun;26(3):9787-9793. PMID 31180311